CLINICAL TRIAL: NCT04599426
Title: Safety and Efficacy of Allogenic NK Cell Transfusion Combined With Azacitidine Therapy for the MDS-EB
Brief Title: Allogenic NK Cell Transfusion Azacitidine MDS-EB
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Second Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020.NK.MDS-EB
Record Dates: First submitted 2020-09-11; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: MDS-EB
Keywords: NK cell MDS-EB

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test Group (Experimental): 10 patients with refractory MDS-RAEB were treated with allogeneic NK cell regimen.
  Interventions: Biological: Allogeneic NK cell regimen group

INTERVENTIONS:
Biological: Allogeneic NK cell regimen group — 10 patients with refractory MDS-RAEB were treated with allogeneic NK cell regimen.
  Allogeneic NK cell regimen ×3 cycle; Cyclophosphamide 300mg/m2.d d1to 3; G-CSF 150ug bid d4-11; Azacitidine 75mg/m2 d5-11; Allogeneic NK cell 10-30×10^6/kg d13，d15 .

SUMMARY:
The aim of this investigation was to assess safety and efficacy of allogenic NK cells therapy for refractory MDS-EB.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with refractory high-risk MDS (MDS-EB1 and EB2) who had no effect of 2 courses of desitabine or CAG or desitabine + CAG.
2. Patients with age 15 years to 70 years.
3. KPS greater than or equal to 60.
4. ALT and AST are less than 3 times normal.
5. Total bilirubin less than 1.5mg/dl(25.65umol/L).
6. Serum creatinine less than 2.5mg/dl(221umol/L), or creatinine scavenging ability greater than or equal to 60 mL/min/1.73 m2.
7. Left ventricular ejection fraction cardiac greater than or equal to 45%, Echocardiography (ECHO) showed no pericardial effusion, Electrocardiogram (ECG) is normal.
8. No pleural effusion in lungs.
9. Oxyhemoglobin saturation greater than or equal to 92% in normal environment.
10. Women of child-bearing age have negative urine pregnancy tests before administration began, and agree to use effective contraception during the trial period up to the last follow-up.
11. KIR mismatch between patient and umbilical cord blood.
12. Volunteer to participate in the trial and sign the informed consent form.

Exclusion Criteria:

1. Malignant tumor patient.
2. Patients who are accompanied by fungal, bacterial, viral, or other uncontrolled infections or require level 4 isolation. (HBV-DNA quantification and normal liver function in patients with hepatitis b infection are excluded).
3. Patients with HIV, HCV positive.
4. Patients with central nervous system diseases, including stroke, epilepsy, dementia, or autoimmune central nervous system disorders.
5. Patients with central nervous system diseases, including stroke, epilepsy, dementia, or autoimmune central nervous system disorders.
6. Patients receiving anticoagulant therapy or with severe coagulation disorders.
7. According to the researcher's judgment, the drug treatment the patient is receiving will affect the safety and effectiveness of the study.
8. Patients with allergies or history of allergies to biological agents used in this program.
9. Lactating or pregnant women.
10. Systemic steroid used within 2 weeks before treatment (except for recent or present use of inhaled corticosteroids).
11. Patients with other uncontrolled diseases, Investigators think it is not suitable for the participants.
12. Any circumstance that the investigator considers may increase the risk to the subject or interfere with the results of the study.
13. Patients participate in other clinical studies.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) (PR+CR) | 3 months
  The proportion of patients with complete response(CR) or partial response(PR) as measured by International Working Group efficacy Criteria for myelodysplastic syndromes

SECONDARY OUTCOMES:
Overall survival(OS) | 1 year
  The proportion of patients with overall survival(OS).

CONTACTS AND LOCATIONS:
Overall Officials: Chengyun Zheng, Ph.D., Study Director — The Second Hospital of Shandong University
Locations (1):
- The 2nd Hospital of Shandong University, Jinan, Shandong, China